CLINICAL TRIAL: NCT00946270
Title: A Phase II, Prospective, Open Label Study (PO-MMM-PI-0011) to Determine the Safety and Efficacy of Pomalidomide (CC-4047) in Subjects With Primary, Post Polycythemia Vera, or Post Essential Thrombocythemia Myelofibrosis (PMF; Post-PV MF, or Post-ET MF)
Brief Title: Pomalidomide for Myelofibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0199; NCI-2012-00360 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Polycythemia Vera; Thrombocythemia
Keywords: CC-4047; Pomalidomide; polycythemia vera; essential thrombocythemia myelofibrosis
MeSH Terms: conditions — Polycythemia Vera; Thrombocytosis | interventions — pomalidomide; Prednisone

STUDY DESIGN:
Intervention Model Description: The first 21 participants received pomalidomide 3.0 mg/day on a 21 day schedule. Due to poor tolerance the study was suspended and amended to treat 20 participants with pomalidomide 0.5 mg/day continuously for 28 days. The study was amended to treat an additional 29 participants with pomalidomide 0.5 mg/day for 28 days plus prednisone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 3 CC-4047 + Prednisone (Experimental): CC-4047 0.5 mg orally daily starting on day 1 through 28. Prednisone given during first 3 cycles of therapy. It will be dosed orally at the dose of 30 mg/day during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
  Interventions: Drug: CC-4047; Drug: Prednisone
- Group 1 CC-4047 (Experimental): CC-4047 3.0 mg orally daily starting on day 1 through 21.
  Interventions: Drug: CC-4047
- Group 2 CC-4047 (Experimental): CC-4047 0.5 mg orally daily starting on day 1 through 28.
  Interventions: Drug: CC-4047

INTERVENTIONS:
Drug: CC-4047 — 0.5 mg capsules daily by mouth day 1 through day 28.
  Other Names: Pomalidomide
  Arms: Group 2 CC-4047; Group 3 CC-4047 + Prednisone
Drug: Prednisone — 30 mg by mouth daily during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
  Arms: Group 3 CC-4047 + Prednisone
Drug: CC-4047 — 3.0 mg capsules daily by mouth day 1 through 21.
  Other Names: Pomalidomide
  Arms: Group 1 CC-4047

SUMMARY:
The goal of this clinical research study is to learn if CC-4047 (now called pomalidomide) and prednisone can help to control MMM. The safety of this therapy will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

CC-4047 is a drug that may also affect the growth of blood vessels that support tumor growth. If these blood vessels stop growing, it may stop cancer cell growth.

Prednisone is a corticosteroid that is similar to a natural hormone made by your body. Prednisone is often given in combination with other chemotherapy to treat cancer.

Study Drug Administration:

On Days 1- 28 of every 28-day study "cycle," you will take CC-4047 capsule(s) by mouth. You should take the capsule(s), about the same time every day. The capsule(s) should not be opened, broken, or chewed. CC-4047 should be taken without food, at least 2 hours before or 2 hours after a meal. If a dose of CC-4047 is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up, rather it should be taken at the next scheduled time point.

In order to take part in this study, you must register into and follow the requirements of the POMALYST REMS™ program of Celgene Corporation. This program provides education and counseling on the risks of exposing unborn children to the study drug, and the risks of blood clots and reduced blood counts. You will be required to receive counseling, follow the pregnancy testing and birth control requirements of the program that are appropriate for you, and take surveys regarding how well you are following with the POMALYST REMS™ program.

You will receive prednisone by mouth during the first 3 cycles of therapy. You will take it 1 time a day during Cycle 1. During Cycle 2, you will take a smaller dose 1 time a day. During Cycle 3, you will take the same dose as in Cycle 2, but only 1 time every other day.

On Days 1-28, you will also take low-dose aspirin. This should be taken at the same time as CC-4047. Aspirin is take to help prevent blood clots, which may occur from taking CC-4047. If you are unable to take aspirin, your study doctor will have you take another drug.

You will be given a study "diary". In this diary, you will record when you take each dose of the study drug. You will return any unused study drug and empty bottles at each visit.

Study Visits:

On Day 1 of Cycles 1 and 2, the following tests and procedures will be performed:

* You will have a physical exam, including measurements of your vital signs (blood pressure, temperature, and heart rate) and weight.
* You will be asked about any drugs you are taking and about recent blood transfusions you may have had.
* You will have a performance status evaluation.
* Blood (about 1 tablespoon) will be drawn for routine tests.

On Days 1, 8, 15, and 22 of Cycles 1 and 2, blood (about 4 teaspoons) will be drawn for routine tests.

On Day 28 of each cycle, the following tests and procedures will be performed:

* You will be asked about any drugs you are taking and about recent blood transfusions you may have had.
* You will be asked about any birth control methods you are using.
* Blood (about 4 tablespoons) will be drawn for routine tests.
* You will be asked about any new side effects or medical conditions you may have experienced.
* You will complete a questionnaire about your quality-of-life as well as an assessment of possible pain in your spleen. (Cycles 1 and 2 only)

On Day 28 of cycles 1,2,3 and every third cycle (Cycle 6, 9, and so on), the following tests and procedures will be performed:

* You will have a physical exam, including measurement of yur vital signs and weight.
* Measurements of your spleen and/or liver will be taken.
* You will have a performance status evaluation.

On Day 28 of every sixth cycle (Cycle 6, 12 and so on)the following tests and procedures will be performed:

* Blood (about 4 teaspoons) will be drawn to test your thyroid function.
* You will have an ECG.
* Response of disease to therapy will be assessed. Bone marrow biopsy and aspirate will be done to confirm a complete response if your doctor thinks it is needed.

Pregnancy Testing:

Women who are able to have children will have a pregnancy test every week during Cycle 1, and then every 28 days after that if your menstrual cycle is regular (If your menstrual cycle is not regular, you will have a blood pregnancy test every 2 weeks). These pregnancy tests will be part of a routine blood draw.

Length of Study:

You will remain on study treatment as long as the therapy is beneficial to you. You will be taken off study early if the disease gets worse or intolerable side effects occur.

End-of-Treatment Visit:

Once you are off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurements of your vital signs and measurements of your spleen and/or liver.
* You will have an ECG.
* You will be asked about any drugs you are taking and about any blood transfusions you may have had.
* Blood (about 4 tablespoons) and urine will be collected for routine tests and thyroid function tests. This routine blood draw will include a pregnancy test for women who are able to have children.
* You will be asked about any side effects you may have experienced.

Follow-Up Visit:

Women who are able to have children will have a blood (about 1 tablespoon) pregnancy test 28 days after the last dose of study drug. If your periods are irregular you will have 2 blood (about 1 tablespoon each time) pregnancy tests, one 14 days after the last dose of study drug and another 28 days after the last dose of study drug. Response of disease to therapy will be assessed at follow-up 28 days after last dose of study drug.

This is an investigational study. CC-4047 (pomalidomide) is FDA approved and commercially available for the treatment of certain types of MM. Its use in this study is investigational.

Prednisone is FDA approved and commercially available.

Up to 70 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Must be >/= 18 years of age at the time of voluntarily signing an Institutional Review Board/Independent Ethics Committee (IRB/IEC) - approved informed consent form.
2. Must be diagnosed with myelofibrosis requiring therapy including myelofibrosis with myeloid metaplasia (MMM), de novo presentation (i.e. agnogenic myeloid metaplasia [AMMM], and developing after an antecedent history of Polycythemia vera (i.e., post-polycythemic myeloid metaplasia [PPMM]), or essential Polycythemia (i.e., post thrombocythemic myeloid metaplasia [PTMM]).
3. Screening total hemoglobin level < 10 g/dL or transfusion-dependent anemia defined as per International Working Group (IWG) criteria (transfusion dependency defined by a history of a least 2 units of red blood cell transfusions in the last 28 days for hemoglobin < 8.5 g/dL that was not associated with overt bleeding)
4. Must have adequate organ function as demonstrated by the following </= 14 days prior to starting study drug: ·Alanine transaminase (ALT) (SGOT) and Aspartate aminotransferase (AST) (SGPT) </= 3 x upper limit of normal (ULN), [unless upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis (EMH)] ·Total bilirubin < 3 x ULN or Direct Bilirubin < 2 x ULN ·Serum creatinine </= 2.5 mg/dL ·Absolute neutrophil count >/= 1,000/µL (>/=1.0 x 10^9/L) ·Platelet count >/= 50,000/µL (>/=50 x 10^9/L)
5. Subjects must be willing to receive transfusion of blood products
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2 at screening.
7. Must be willing to adhere to the study visit schedule and other protocol requirements.
8. No active malignancies with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma (in situ) of the cervix or breast
9. All study participants must be registered into the mandatory POMALYST REMS™ program, and be willing and able to comply with the requirements of the POMALYST REMS™ program.
10. Females of reproductive potential (FCBP†) must adhere to the scheduled pregnancy testing as required in the POMALYST REMS™ program. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Known positive status for HIV, hepatitis B carrier, or active hepatitis C infection.
2. The use of any growth factors, cytotoxic chemotherapeutic agents (e.g. hydroxyurea), corticosteroids, or experimental drug or therapy within 14 days of starting CC-4047 and/or lack of recovery from all toxicity from previous therapy to grade 1 or better.
3. Any serious medical condition or psychiatric illness that would prevent, (as judged by the treating physician) the subject from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Pregnant or lactating females
5. Prior use of CC-4047
6. Currently enrolled on another clinical trial or receiving investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-07-22 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Daver N, Shastri A, Kadia T, Newberry K, Pemmaraju N, Jabbour E, Zhou L, Pierce S, Cortes J, Kantarjian H, Verstovsek S. Phase II study of pomalidomide in combination with prednisone in patients with myelofibrosis and significant anemia. Leuk Res. 2014 Sep;38(9):1126-9. doi: 10.1016/j.leukres.2014.06.015. Epub 2014 Jul 6. PMID 25047979
- [Derived] Daver N, Shastri A, Kadia T, Quintas-Cardama A, Jabbour E, Konopleva M, O'Brien S, Pierce S, Zhou L, Cortes J, Kantarjian H, Verstovsek S. Modest activity of pomalidomide in patients with myelofibrosis and significant anemia. Leuk Res. 2013 Nov;37(11):1440-4. doi: 10.1016/j.leukres.2013.07.007. Epub 2013 Jul 25. PMID 23890523
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 2009 to March 2013.
Groups:
- Group 1: Oral CC-4047 3.0 mg: CC-4047 3.0 mg orally daily.
  CC-4047: 3.0 mg orally daily starting on day 1 through 21.
- Group 2: Oral CC-4047 0.5 mg: CC-4047 0.5 mg orally daily .
  CC-4047: 0.5 mg orally daily starting on day 1 through 28.
- Group 3: Oral CC-4047 0.5 mg + Prednisone: CC-4047 0.5 mg orally daily. Prednisone given during first 3 cycles of therapy. It will be dosed orally at the dose of 30 mg/day during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
  CC-4047: 0.5 mg capsules daily by mouth day 1 through day 28.
  Prednisone: 30 mg by mouth daily during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
Period: Overall Study
Arm/Group | Group 1: Oral CC-4047 3.0 mg | Group 2: Oral CC-4047 0.5 mg | Group 3: Oral CC-4047 0.5 mg + Prednisone
Started | 21 | 20 | 29
Completed | 21 | 20 | 29
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 3 CC-4047 + Predniaone: CC-4047 0.5 mg orally daily. Prednisone given during first 3 cycles of therapy. It will be dosed orally at the dose of 30 mg/day during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
  CC-4047: 0.5 mg capsules daily by mouth day 1 through day 28.
  Prednisone: 30 mg by mouth daily during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
- Total: Total of all reporting groups
Arm/Group | Group 1 CC-4047 | Group 2 CC-4047 | Group 3 CC-4047 + Predniaone | Total
Number analyzed (Participants) | 21 | 20 | 29 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 8 | 25
  >=65 years | 11 | 13 | 21 | 45
Age, Continuous [Median (Full Range); unit: years] | 66 [53 to 82] | 69 [39 to 86] | 69 [48 to 88] | 68 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 29
  Male | 11 | 10 | 20 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 1 | 7
  White | 19 | 15 | 28 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 29 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Overall Response
Description: Primary endpoint is best overall response. An evaluable subject classified as a treatment success for the primary endpoint if the subject's best overall response is clinical improvement (CI) as determined by International Working Group Criteria over the first 6 cycles of study treatment. International Working Group (IWG) consensus criteria for treatment response in myelofibrosis - Clinical improvement (CI) in anemia 1/ A minimum 20g/L increase in hemoglobin level or 2. becoming transfusion independent for at least 8 week duration.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: CC-4047 0.5 mg orally daily starting on day 1 through 28.
- Group 3 CC-4047 + Prednisone: CC-4047 0.5 mg orally daily. Prednisone given during first 3 cycles of therapy. It will be dosed orally at the dose of 30 mg/day during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
  CC-4047: 0.5 mg capsules daily by mouth day 1 through day 28.
  Prednisone: 30 mg by mouth daily during cycle 1, 15 mg/day during cycle 2, and 15 mg every other day during cycle 3, and then it will be discontinued.
Arm/Group | Group 1 CC-4047 | Group 2 | Group 3 CC-4047 + Prednisone
Number analyzed (Participants) | 21 | 20 | 29
Participants | 0 | 3 | 6

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Group 1 CC-4047 | Group 2 CC-4047 | Group 3 CC-4047 + Prednisone
All-Cause Mortality (participants affected / at risk) | 2/21 | 3/20 | 1/29
Serious Adverse Events (participants affected / at risk) | 15/21 | 8/20 | 11/29
Other Adverse Events (participants affected / at risk) | 13/21 | 10/20 | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 CC-4047 (N=21) | Group 2 CC-4047 (N=20) | Group 3 CC-4047 + Prednisone (N=29)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 1 (4) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (4) | 1 (2)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device Complication (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Edema Limb (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fistula Rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid Overload - post transfusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (4)
Intra-operative injury (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (8) | 0 (0) | 0 (0)
Neutropenic Fever (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Peripheral Edema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Pneumonitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Pulmonary Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rigors/Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic infarct (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Stricture/Stenosis Esophagus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Subdural Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 CC-4047 (N=21) | Group 2 CC-4047 (N=20) | Group 3 CC-4047 + Prednisone (N=29)
Abdominal hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac general (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascualr Ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspena (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fall (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (2)
Abnormal Gait (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Iron increased (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT00946270/Prot_SAP_000.pdf